CLINICAL TRIAL: NCT01185821
Title: A Dose Blinded Extension Study to the CBAF312A2201 Study to Evaluate Long-term Safety, Tolerability and Efficacy of BAF312 Given Orally Once Daily in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Long-term Safety, Tolerability and Efficacy of BAF312 Given Orally in Patients With Relapsing-remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBAF312A2201E1; 2009-014392-51 (EudraCT Number)
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: BAF312; siponimod; Multiple Sclerosis; Relapsing remitting Multiple Sclerosis; Demyelinating Autoimmune Diseases; MS; RRMS; inflammatory disease
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — siponimod

STUDY DESIGN:
Intervention Model Description: This extension study was originally set up as a 2 year dose-blinded extension study to maintain blinding of ongoing Core study. Study was later amended to include a subsequent Open-Label treatment phase after Core study was unblinded. During the Dose-Blinded phase of the extension study patients received the same dose from the Core study. Patients who received placebo in Period 1 during the Core Study were equally randomized to 1 of the 3 active doses of siponimod used during Period 1 (0.5, 2.0, or 10 mg) and patients who received placebo in Period 2 were equally randomized to 1 of the 2 active doses of siponimod used during Period 2 (0.25 mg or 1.25 mg).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking continued during the double blind period of extension only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BAF312 10 mg/2 mg (Experimental): 10 mg dose in Double Blind Phase and 2 mg in Open Label Phase
  Interventions: Drug: BAF312
- BAF312 2 mg/2 mg (Experimental): 2 mg dose in Double Blind Phase and 2 mg in Open Label Phase
  Interventions: Drug: BAF312
- BAF312 1.25 mg/2 mg (Experimental): 1.25 mg dose in Double Blind Phase and 2 mg in Open Label Phase
  Interventions: Drug: BAF312
- BAF312 .5 mg/2 mg (Experimental): .5 mg dose in Double Blind Phase and 2 mg in Open Label Phase
  Interventions: Drug: BAF312
- BAF312 .25 mg/2 mg (Experimental): .25 mg dose in Double Blind Phase and 2 mg in Open Label Phase
  Interventions: Drug: BAF312

INTERVENTIONS:
Drug: BAF312 — BAF312 was supplied in film-coated tablets in strengths of 5, 4 ,2, 1, .5 and .25 mg. The actual doses taken were 10, 2, 1.25, .5 and .25 mg taken orally once a day.
  Other Names: siponimod

SUMMARY:
This study consisted of a two year dose blinded phase during which patients received one of five doses of siponimod (10, 2, 1.25, 0.5 or 0.25mg) following which patients were switched to open label treatment with siponimod 2mg for approximately a further 3 years. It will provide data on long term safety, tolerability and efficacy of siponimod in the RRMS patient population

DETAILED DESCRIPTION:
This study was prematurely discontinued after approximately 5 years. The decision to prematurely discontinue the study was not taken due to safety-related concerns, rather due to a decision to focus the development of siponimod in MS on a different population.

ELIGIBILITY:
Inclusion Criteria:

* Patients completed the core study BAF312A2201
* Written informed consent provided before any assessment of the extension study
* Female patients at risk of becoming pregnant must have a negative pregnancy test and use simultaneously two forms of effective contraception

Exclusion Criteria:

* Newly diagnosed systemic disease other than MS (which may require immunosuppressive treatment)
* Malignancies, diabetes, significant cardiovascular and pulmonary diseases and conditions
* Active infections

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2010-08-30 (Actual); Primary Completion 2016-10-10 (Actual); Study Completion 2016-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (42):
- United States (8):
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Pompano Beach, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Grand Rapids, Michigan
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Seattle, Washington
- Canada (3):
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Gatineau, Quebec
  - Novartis Investigative Site, Greenfield Park, Quebec
- Finland (2):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Tampere
- Germany (4):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Ibbenbueren
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Veszprém
- Italy (3):
  - Novartis Investigative Site, Montichiari, BS
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Roma, RM
- Norway (2):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo
- Poland (3):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
- Russia (3):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (3):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Zurich
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Haseki / Istanbul
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli

REFERENCES:
- [Derived] Kappos L, Li DK, Stuve O, Hartung HP, Freedman MS, Hemmer B, Rieckmann P, Montalban X, Ziemssen T, Hunter B, Arnould S, Wallstrom E, Selmaj K. Safety and Efficacy of Siponimod (BAF312) in Patients With Relapsing-Remitting Multiple Sclerosis: Dose-Blinded, Randomized Extension of the Phase 2 BOLD Study. JAMA Neurol. 2016 Sep 1;73(9):1089-98. doi: 10.1001/jamaneurol.2016.1451. PMID 27380540

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients enrolled in the Extension study had completed the Core study. All patients underwent a 10 day titration at the start of the dose blinded phase of the study
Pre-assignment Details: During the double blind phase of the extension study patients received the same dose from the Core study. Placebo patients from Core Period 1 were randomized to 0.5, 2 or 10mg, those from Period 2 were randomized to 0.25 or 1.25 mg. All patients received 2mg in Open Label phase (.5 and .25mg were titrated up to 2mg)
Period: Overall Study
Arm/Group | BAF312 10 mg/2 mg | BAF312 2 mg/2 mg | BAF312 1.25 mg/2 mg | BAF312 .5 mg/2 mg | BAF312 .25 mg/2 mg
Started | 33 | 29 | 43 | 29 | 50
Patients With Washout | 33 | 29 | 39 | 29 | 33
Patients Without Washout | 0 | 0 | 4 | 0 | 17
Patients on Placebo in Core | 8 | 7 | 9 | 8 | 2
Completed | 26 | 20 | 33 | 23 | 26
Not Completed | 7 | 9 | 10 | 6 | 24
Not completed — Abnormal laboratory value(s) | 1 | 2 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 1
Not completed — Abnormal test procedure result | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Condition no longer required study drug | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 2 | 3 | 1 | 2 | 5
Not completed — Lack of Efficacy | 0 | 0 | 3 | 0 | 9
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 1 | 3
Not completed — Lost to Follow-up | 1 | 1 | 2 | 1 | 2
Not completed — Administrative problems | 0 | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Extension set consisted of all patients who received at least one dose of Extension study drug who do not have a major protocol deviation.
Groups:
- Total: Total of all reporting groups
Arm/Group | BAF312 10 mg/2 mg | BAF312 2 mg/2 mg | BAF312 1.25 mg/2 mg | BAF312 .5 mg/2 mg | BAF312 .25 mg/2 mg | Total
Number analyzed (Participants) | 33 | 29 | 43 | 29 | 50 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (9.09) | 35.1 (9.16) | 34.0 (7.57) | 35.2 (9.10) | 37.2 (8.42) | 35.7 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 32 | 18 | 41 | 130
  Male | 12 | 11 | 11 | 11 | 9 | 54
Expanded disability status scale (EDSS) [Mean (Standard Deviation); unit: units on a scale] — Disability progression was assessed based on the EDSS scores ranging from 0 (normal) to 10 (death due to MS)
  units on a scale | 2.03 (0.960) | 2.19 (1.278) | 1.95 (1.096) | 1.88 (1.374) | 2.22 (1.258) | 2.07 (1.190)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Adverse Events During Evaluation of Long Term Safety and Tolerability of BAF312A in Extension Study.
Description: Refer to adverse events for complete listing of serious adverse events and other adverse events. Adverse events of interest were presented in separate tables. There were no reports of macular edema.
Time Frame: Baseline up to approximately 5 years
Measure: Number; unit: events
Arm/Group | BAF312 10 mg/2 mg | BAF312 2 mg/2 mg | BAF312 1.25 mg/2 mg | BAF312 .5 mg/2 mg | BAF312 .25 mg/2 mg
Number analyzed (Participants) | 33 | 29 | 43 | 29 | 50
events
  Serious adverse events | 4 | 7 | 6 | 6 | 8
  Other adverse events | 30 | 26 | 42 | 29 | 42

2. Primary Outcome: Number of Participants With Cardiac Conduction Abnormalities During the Titration Phase of the Study (Without Washout)
Description: Number of patients with abnormal ECG conduction findings during dose-blinded titration at any visit post-dose, by type of abnormality and treatment (Extension Set). Number analyzed represent participants who had ECG results. Washout was defined as not being on treatment drug between Core and Extension for >7 days. Abbreviation: Con=conduction, IVCD=intraventricular conduction defect , WPW=Wolff-Parkinson-White syndrome
Time Frame: Baseline Extension up to day 10
Measure: Number; unit: participants
Arm/Group | BAF312 10 mg/2 mg | BAF312 2 mg/2 mg | BAF312 1.25 mg/2 mg | BAF312 .5 mg/2 mg | BAF312 .25 mg/2 mg
Number analyzed (Participants) | 33 | 29 | 39 | 29 | 33
participants
  Conduction-Prolonged QTc | 5 | 2 | 5 | 2 | 4
  Conduction - IVCD | 3 | 8 | 1 | 3 | 0
  Conduction - AV Mobitz I | 1 | 0 | 0 | 0 | 0
  Con:1st degree AV block | 0 | 1 | 1 | 1 | 1
  Conduction - WPW | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With Cardiac Conduction-IVCD Abnormality During the Titration Phase of the Study (With Washout)
Description: Number of patients with abnormal ECG conduction findings during dose-blinded titration at any visit post-dose, by type of abnormality and treatment (Extension Set). Number analyzed represent participants who had ECG results. Washout was defined as not being on treatment drug between Core and Extension for >7 days. Abbreviations: washout = WO, Con=conduction
Time Frame: Baseline Extension up to day 10
Measure: Number; unit: participants
Arm/Group | BAF312 .25 mg/2 mg
Number analyzed (Participants) | 4
participants | 4

4. Primary Outcome: Number of Participants With Changes in Blood Pressure for Overall Extension Study. (Extension Analysis Set)
Description: Sitting blood pressure was measured in triplicate. The categories of notably low and high values and changes are presented for systolic (SBP) and diastolic (DBP). Multiple occurrences for a patient are counted as one occurrence in this table.
Time Frame: Baseline Extension up to approximately 5 years
Measure: Number; unit: participants
Arm/Group | BAF312 10 mg/2 mg | BAF312 2 mg/2 mg | BAF312 1.25 mg/2 mg | BAF312 .5 mg/2 mg | BAF312 .25 mg/2 mg
Number analyzed (Participants) | 33 | 29 | 43 | 29 | 50
participants
  SBP Low: ≤ 90 | 1 | 3 | 2 | 1 | 1
  SBP ≥ 20 decrease from baseline | 8 | 10 | 4 | 6 | 10
  SBP High: ≥ 160 | 1 | 1 | 1 | 3 | 3
  SBP ≥ 20 increase from baseline | 9 | 8 | 12 | 13 | 18
  DBP Low: ≤ 50 | 1 | 0 | 1 | 0 | 1
  DBP ≥ 15 decrease from baseline | 14 | 8 | 10 | 10 | 10
  DBP High: ≥ 100 | 4 | 7 | 4 | 4 | 4
  DBP ≥ 15 increase from baseline | 9 | 13 | 13 | 11 | 17

5. Primary Outcome: Number of Participants With Viral Infections of Interest Greater or Equal to 5% in Any Dose Group (Extension Set)
Description: Most infections were clinical diagnoses and were not confirmed by microbiology / virologic investigations. A patient with multiple occurrences of an infection for a preferred term is counted only once in each specific category.
  Events identified as infections by the Investigator and defined as an AE with onset on or after the first dose of Extension Study drug up to and including 30 days after the date of the last dose
Time Frame: Baseline Extension up to approximately 5 years
Measure: Number; unit: participants
Arm/Group | BAF312 10 mg/2 mg | BAF312 2 mg/2 mg | BAF312 1.25 mg/2 mg | BAF312 .5 mg/2 mg | BAF312 .25 mg/2 mg
Number analyzed (Participants) | 33 | 29 | 43 | 29 | 50
participants
  Oral herpes | 5 | 0 | 4 | 2 | 4
  Herpes zoster | 5 | 0 | 3 | 2 | 0
  Influenza | 3 | 4 | 3 | 6 | 6

6. Primary Outcome: Number of Participants With Dermatologic Alterations - Basal Cell Carcinoma (Extension Set)
Time Frame: Baseline Extension up to approximately 5 years
Measure: Number; unit: participants
Arm/Group | BAF312 10 mg/2 mg | BAF312 2 mg/2 mg | BAF312 1.25 mg/2 mg | BAF312 .5 mg/2 mg | BAF312 .25 mg/2 mg
Number analyzed (Participants) | 33 | 29 | 43 | 29 | 50
participants | 1 | 0 | 1 | 0 | 1

7. Secondary Outcome: Number of Relapses in One Year - Annualized Relapse Rates for Overall Extension Study (ARR) (Extension Set)
Description: Group level ARR (raw) is calculated as the total number of relapses for all the patients in the treatment group divided by the total number of days on study for all patients in the group and multiplied by 365.25 to obtain the annual rate.
  Model estimates are based on a negative binomial regression model, adjusted for treatment group, age, baseline EDSS, baseline number of Gd-enhanced T1 lesions and number of relapses in previous 2 years as covariates, with log(time on study in years) as the offset variable, using the log link.
Time Frame: Baseline extension up to approximately 5 years
Measure: Mean (95% Confidence Interval); unit: Group level ARR
Arm/Group | BAF312 10 mg/2 mg | BAF312 2 mg/2 mg | BAF312 1.25 mg/2 mg | BAF312 .5 mg/2 mg | BAF312 .25 mg/2 mg
Number analyzed (Participants) | 33 | 29 | 43 | 29 | 50
Group level ARR | 0.18 [0.11 to 0.31] | 0.15 [0.08 to 0.26] | 0.16 [0.10 to 0.26] | 0.19 [0.11 to 0.33] | 0.22 [0.14 to 0.35]

8. Secondary Outcome: Percentage of Participants Free of Magnetic Resonance Imaging (MRI) Identified Disease Activity at Any Scan During Extension Study (Extension Set)
Description: Free of MRI disease activity is defined as free of Gadolinium enhanced T1 lesions at any scan; free of new or enlarging T2 lesions at any scan: free of both gadolinium enhanced T1 lesions and new or enlarging T2 lesions at any scan. Number of patients analyzed = patients with at least one MRI scan during the specified time period. New lesions at a specific visit are assessed relative to the previous scheduled visit scan.
  No imputation of missing scans is performed. As a result missing scans can lead to an overestimation of the proportion of patients free of a specific MRI activity.
Time Frame: Baseline Extension up to approximately 5 years
Measure: Number; unit: percentage of participants
Arm/Group | BAF312 10 mg/2 mg | BAF312 2 mg/2 mg | BAF312 1.25 mg/2 mg | BAF312 .5 mg/2 mg | BAF312 .25 mg/2 mg
Number analyzed (Participants) | 31 | 26 | 43 | 29 | 47
percentage of participants
  Free of Gd-enhanced T1 lesions at any scan | 58.1 | 57.7 | 58.1 | 44.8 | 66.0
  Free of new/enlarging T2 lesions at any scan | 32.3 | 42.3 | 46.5 | 20.7 | 40.4
  Free of Gd-enhanced T1 and new enlarged T2 lesions | 32.3 | 42.3 | 44.2 | 20.7 | 40.4

9. Secondary Outcome: Percentage of Participants Free of Confirmed Disability Progression in Extension Study (Extension Set)
Description: Six-month disability progression was defined relative to extension baseline EDSS score: 1.5 point increase in patients with baseline EDSS score of 0, 1.0 increase in patients with baseline EDSS score of between 0.5 to 5.0, inclusive and 0.5 increase in patients with baseline EDSS score of ≥ 5.5. The criteria for 6-month disability progression included detection of onset of progression and confirmation of progression for a period of at least 6 months.
Time Frame: Baseline Extension up to approximately 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BAF312 10 mg/2 mg | BAF312 2 mg/2 mg | BAF312 1.25 mg/2 mg | BAF312 .5 mg/2 mg | BAF312 .25 mg/2 mg
Number analyzed (Participants) | 33 | 29 | 43 | 29 | 50
percentage of participants | 72.3 [56.0 to 88.7] | 82.4 [66.6 to 98.3] | 84.8 [73.5 to 96.0] | 81.4 [66.6 to 96.1] | 78.6 [65.4 to 91.9]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV)until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Groups:
- BAF312 10/2 mg: BAF312 10/2 mg
- BAF312 2/2 mg: BAF312 2/2 mg
- BAF312 1.25/2 mg: BAF312 1.25/2 mg
- BAF312 0.5/2 mg: BAF312 0.5/2 mg
- BAF312 0.25/2 mg: BAF312 0.25/2 mg
- All Patients: All patients
Arm/Group | BAF312 10/2 mg | BAF312 2/2 mg | BAF312 1.25/2 mg | BAF312 0.5/2 mg | BAF312 0.25/2 mg | All Patients
Serious Adverse Events (participants affected / at risk) | 4/33 | 7/29 | 6/43 | 6/29 | 8/50 | 31/184
Other Adverse Events (participants affected / at risk) | 30/33 | 26/29 | 42/43 | 29/29 | 42/50 | 169/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BAF312 10/2 mg (N=33) | BAF312 2/2 mg (N=29) | BAF312 1.25/2 mg (N=43) | BAF312 0.5/2 mg (N=29) | BAF312 0.25/2 mg (N=50) | All Patients (N=184)
Splenic cyst (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Otosclerosis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Submandibular mass (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Smear cervix abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 3
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Drug abuse (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1
Uterine cervical metaplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3.999% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BAF312 10/2 mg (N=33) | BAF312 2/2 mg (N=29) | BAF312 1.25/2 mg (N=43) | BAF312 0.5/2 mg (N=29) | BAF312 0.25/2 mg (N=50) | All Patients (N=184)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2 | 0 | 3
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 2
Lymphopenia (Blood and lymphatic system disorders) | 6 | 5 | 4 | 6 | 3 | 24
Palpitations (Cardiac disorders) | 0 | 2 | 0 | 0 | 1 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 2 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 2 | 0 | 1 | 4
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 2 | 3
Vertigo (Ear and labyrinth disorders) | 4 | 1 | 3 | 2 | 6 | 16
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 1 | 3
Conjunctivitis (Eye disorders) | 1 | 0 | 2 | 1 | 1 | 5
Eye pain (Eye disorders) | 2 | 0 | 0 | 1 | 0 | 3
Iridocyclitis (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 2
Vision blurred (Eye disorders) | 2 | 0 | 3 | 0 | 0 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 3 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 3 | 5 | 3 | 12
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 7 | 3 | 6 | 19
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2 | 5
Enteritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 1 | 6
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 4 | 8
Toothache (Gastrointestinal disorders) | 0 | 2 | 4 | 1 | 4 | 11
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 3 | 7
Asthenia (General disorders) | 0 | 1 | 2 | 0 | 1 | 4
Fatigue (General disorders) | 1 | 4 | 5 | 2 | 6 | 18
Gait disturbance (General disorders) | 3 | 0 | 0 | 1 | 0 | 4
Influenza like illness (General disorders) | 1 | 0 | 2 | 1 | 1 | 5
Non-cardiac chest pain (General disorders) | 3 | 0 | 1 | 0 | 2 | 6
Oedema peripheral (General disorders) | 0 | 2 | 0 | 1 | 0 | 3
Pyrexia (General disorders) | 2 | 1 | 4 | 3 | 5 | 15
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 3
Bronchitis (Infections and infestations) | 0 | 2 | 5 | 3 | 6 | 16
Conjunctivitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 3
Cystitis (Infections and infestations) | 3 | 1 | 2 | 1 | 1 | 8
Fungal infection (Infections and infestations) | 3 | 1 | 0 | 1 | 1 | 6
Fungal skin infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 2 | 1 | 3 | 4 | 10
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 3 | 0 | 2 | 5
Herpes zoster (Infections and infestations) | 5 | 0 | 3 | 2 | 0 | 10
Influenza (Infections and infestations) | 4 | 4 | 5 | 7 | 7 | 27
Nasopharyngitis (Infections and infestations) | 10 | 8 | 17 | 11 | 18 | 64
Onychomycosis (Infections and infestations) | 1 | 1 | 0 | 0 | 3 | 5
Oral herpes (Infections and infestations) | 5 | 0 | 4 | 2 | 4 | 15
Otitis media (Infections and infestations) | 1 | 1 | 0 | 0 | 3 | 5
Pharyngitis (Infections and infestations) | 1 | 4 | 3 | 6 | 3 | 17
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 4
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 2 | 5
Rhinitis (Infections and infestations) | 3 | 2 | 1 | 0 | 1 | 7
Sinusitis (Infections and infestations) | 3 | 2 | 3 | 5 | 5 | 18
Subcutaneous abscess (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 2
Tinea versicolour (Infections and infestations) | 0 | 2 | 2 | 0 | 1 | 5
Tonsillitis (Infections and infestations) | 1 | 1 | 5 | 2 | 1 | 10
Tooth infection (Infections and infestations) | 1 | 2 | 1 | 1 | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 4 | 7 | 9 | 30
Urinary tract infection (Infections and infestations) | 6 | 4 | 2 | 4 | 4 | 20
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 2 | 2 | 5
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | 4
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 3 | 1 | 8
Fall (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 2 | 1 | 9
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 2 | 1 | 7
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 3
Alanine aminotransferase increased (Investigations) | 3 | 5 | 3 | 2 | 2 | 15
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 2
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 2 | 1 | 4
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 0 | 3 | 5
Gamma-glutamyltransferase increased (Investigations) | 3 | 3 | 2 | 3 | 2 | 13
Hepatic enzyme increased (Investigations) | 2 | 1 | 1 | 0 | 1 | 5
Lymphocyte count decreased (Investigations) | 4 | 2 | 4 | 2 | 3 | 15
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 4 | 2 | 1 | 3 | 12
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 2 | 3 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 5 | 3 | 3 | 19
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 1 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 0 | 2 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 4 | 5 | 12
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 2 | 6
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 1 | 0 | 5
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 6 | 2 | 7 | 18
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 4 | 7
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 1 | 2 | 2 | 10
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1 | 0 | 3
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 1 | 4 | 8
Headache (Nervous system disorders) | 9 | 4 | 9 | 4 | 10 | 36
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 2 | 4
Migraine (Nervous system disorders) | 2 | 0 | 3 | 1 | 0 | 6
Muscle spasticity (Nervous system disorders) | 0 | 2 | 0 | 3 | 0 | 5
Neuralgia (Nervous system disorders) | 1 | 0 | 4 | 0 | 0 | 5
Paraesthesia (Nervous system disorders) | 4 | 0 | 0 | 2 | 3 | 9
Anxiety (Psychiatric disorders) | 3 | 1 | 1 | 0 | 4 | 9
Depression (Psychiatric disorders) | 1 | 1 | 6 | 3 | 7 | 18
Insomnia (Psychiatric disorders) | 1 | 2 | 8 | 3 | 6 | 20
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0 | 3
Bladder dysfunction (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 2
Micturition urgency (Renal and urinary disorders) | 2 | 1 | 1 | 0 | 1 | 5
Nephrolithiasis (Renal and urinary disorders) | 2 | 2 | 0 | 1 | 0 | 5
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0 | 3
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3 | 4 | 2 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 0 | 3 | 10
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 1 | 5
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 0 | 1 | 8
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 2
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 3 | 7
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1 | 1 | 5
Hypertension (Vascular disorders) | 1 | 1 | 3 | 3 | 8 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.